CLINICAL TRIAL: NCT03754946
Title: The Critical Threshold of Pulse Oximetry Plethysmographic Waveform Parameters in High Quality CPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201502019
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: cardiopulmonary resuscitation; pulse oximetry plethysmographic waveform; quality monitor; partial pressure of end-tidal carbon dioxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to analyze the relationship of the area under the curve (AUC) and/or the amplitude (Amp) of pulse oximetry plethysmographic waveform (POP) with partial pressure of end-tidal carbon dioxide (PETCO2) which could be used to reflect its quality in cardiopulmonary resuscitation (CPR), and then to determine the critical threshold of POP parameters in high quality CPR.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrested
* The time from cardiac arrest to receiving basic life support is less than 10 minutes
* Get advanced life support (endotracheal intubation and PETCO2 monitoring)

Exclusion Criteria:

* Defuse CPR
* chronic obstructive pulmonary disease (COPD) with type II respiratory failure
* Terminal malignant tumors or terminal stage of other diseases
* Rib fracture
* Cardiac arrest caused by hemorrhagic shock pulmonary embolism and cardiac tamponade
* Sever anemia(HGB<7g/dl)
* Untreated tension pneumothorax
* Tinea unguium, dyeing Fingernails and other factors affect the monitor of Pulse Oximetry Plethysmographic Waveform such vasculitis and Raynaud's phenomenon

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the participant hospitals and met the inclusion criteria were included in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
the cut-off value of POP parameters in High Quality CPR | one year
  Describe the the cut-off value of POP parameters in High Quality CPR. Receiver operating curve analysis was performed to evaluate the accuracy in predicting return of spontaneous circulation (ROSC).
Compare different predictors | one year
  Area under curve (AUC) between potential predictors was compared by using a nonparametric test, and the optimal cutoff point was determined by estimating the Youden's index.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China